CLINICAL TRIAL: NCT04937621
Title: Study of Arrhythmia and ECG Abnormalities in Patients With COVID-19
Acronym: RYTHMO-COV
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/18
Record Dates: First submitted 2021-06-22; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Arrhythmia; SARS-CoV-2 Infection
Keywords: COVID-19; ECG; Torsade de pointe; QT interval
MeSH Terms: conditions — Arrhythmias, Cardiac; COVID-19; Torsades de Pointes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 infection: This group includes patients prospectively included during their follow-up at the Bordeaux University Hospital for COVID-19, as well as retrospectively included patients whose follow-up for COVID-19 has been completed.
  Interventions: Diagnostic Test: ECG data analysis; Drug: Treatment data collect; Biological: Biological check-up data collect; Other: Collection of clinical events of interest

INTERVENTIONS:
Diagnostic Test: ECG data analysis — Baseline ECG as well as follow-up ECG are analysed
Drug: Treatment data collect — Baseline treatment data as well as follow-up treatment data are collected
Biological: Biological check-up data collect — Baseline Biological check-up data as well as follow-up data are collected
Other: Collection of clinical events of interest — Clinical events of interest at the baseline as well as follow-up clinical events are collected

SUMMARY:
Cardiac involvement has been described in Severe Acute Respiratory Syndrome - Coronavirus-2 (SARS-CoV-2) infection. Although there are no approved drugs to prevent or treat SARS-CoV-2 infection at present time, several medications used have the potential to increase QT interval and eventually provoke torsades de pointe. The investigators therefore create a study that include all patients with SARS-CoV-2 infection having an electrocardiogram (ECG). The investigators evaluate the percentage of patients with ECG abnormalities, describe the abnormalities and evaluate the occurrence of syncope, ventricular arrhythmia and corrected QT (cQT) interval modification in patients receiving treatment.

DETAILED DESCRIPTION:
In patients with SARS-CoV-2 infection, the investigators analyze baseline ECG as well as follow-up ECG. Patients followed by Bordeaux University Hospital for COVID-19 can be included. ECG are digitized in the computerized patient file (DxCARE) for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of both gender,
* Followed by Bordeaux University Hospital for SARS-CoV-2 infection with a cardiac monitoring or ECG realized.
* Non opposition expressed.

Exclusion Criteria:

* Minor,
* Inability to understand the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with SARS-CoV-2 infection followed by Bordeaux University Hospital for COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of ECGs abnormalities in patients SARS-CoV-2 infection | Day 0
  Percentage of ECGs with abnormalities

SECONDARY OUTCOMES:
Evolution of PR, QRS and cQT interval | Baseline and 1 month
  The evolution of interval is measured in seconds for patients receiving drugs interfering with cardiac electrophysiology for SARS-CoV-2 infection
Rate of syncope during treatment | Baseline and 1 month
  The number of syncope is measured during the treatment
Rate of cardiac death during treatment | Baseline and 1 month
  The number of cardiac death is measured during the treatment
Rate of arrhythmia during treatment | Baseline and 1 month
  The number of arrhythmia is measured during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: frédéric Sacher, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France

IPD SHARING:
Plan to Share IPD: No